CLINICAL TRIAL: NCT04019886
Title: Impact of Neurophysiological Facilitation of Respiration in Preterm Neonates Admitted in Level II Neonatal Intensive Care Unit: A Randomized Controlled Trail
Brief Title: Impact of Neurophysiological Facilitation of Respiration in Preterm Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDU/IEC/2019/03
Record Dates: First submitted 2019-07-02; First posted 2019-07-15 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: Preterm; Neonates; Neurofacilitation Technique; Respiration
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): It consists following techniques-
  1. Peri-oral stimulation
  2. Vertebral pressure
  3. Anterior stretch -lifting posterior basal area
  4. Co-contraction -abdomen
  5. Intercoastal stretch
  6. Moderate manual pressure
  Interventions: Other: Neurophysiological Facilitation of Respiration
- Control Group (No Intervention): Outcome measure will be measured at baseline on first day prior to the intervention and on 5th day after the treatment.

INTERVENTIONS:
Other: Neurophysiological Facilitation of Respiration — Six neuro-facilitation techniques will be given to experimental group. Each technique will be given for 5 seconds hold with 5 repetitions and two sets.
  Arms: Experimental Group

SUMMARY:
Background: Respiratory distress syndrome (RDS) or Neonatal respiratory distress syndrome (NRDS) is characterized by pulmonary insufficiency, in preterm neonates and is the major cause of death in preterm. Neurophysiological facilitation of Respiration (NFR) technique produce reflex respiratory movement response, as it involves application of external proprioceptive and tactile stimuli that is known to alter the rate and depth of breathing Aim: This study is being conducted to determine the effectiveness of NFR in preterm neonates diagnosed with RDS.

Methods: In this study 30 preterm (1- 8 days) neonates diagnosed with Respiratory Distress Syndrome will be taken and assigned into two groups,Experimental group (n=15) and control group (n=15). Neonates within eight days of birth those born before 37 weeks of gestation, diagnosed with RDS were included in the study. Neonate undergone recent surgery or congenital disorder, or medically unstable will be excluded.

Data analysis: Normality of the collected data will be analyzed with either two of the normality test i.e. Shapiro Wilk test and Kolmogorov Smirnov test based on sample size. Demographics characteristic of collected sample will be expressed in a mean standard deviation or median and range based normality. For Between group comparison Independent t test or Mann Whitney U test and for within group comparison paired t test or Wilcoxon singed ranked test will be used.

DETAILED DESCRIPTION:
1. Introduction:

   Respiratory distress syndrome (RDS) or Neonatal respiratory distress syndrome (NRDS) is characterized by pulmonary insufficiency, in preterm neonates and is the major cause of death in preterm. The major cause of RDS is surfactant deficiency. Main features of respiratory distress syndrome are retraction, grunting and tachypnoea and sometimes cyanosis is also present as an associated sign.There are various types of Physiotherapy Interventions given for respiratory disorders in neonates, namely they are chest percussion, vibration and shaking, postural drainage (gravity assisted), Neurophysiological Facilitation of Respiration (NFR). NFR technique produce reflex respiratory movement response, as it involves application of external proprioceptive and tactile stimuli that is known to alter the rate and depth of breathing.

   1.1Problem statement: Role of pulmonary NFR has shown to be effective in adult patients with COPD and in geriatric population. This study aims to evaluate the effectiveness of NFR in neonates with respiratory conditions.

   1.2 Objective of the study: To demonstrate the benefit of NFR in hospitalised neonates with Respiratory Distress Syndrome (RDS).
2. Procedure:

Participants will be selected by simple random sampling method according to the selection criteria.Procedure will be explained to the patient and written consent will be taken from them.

Outcome measures will be taken on the first day prior to the intervention and on the 5th day after the intervention. Outcome measure used will be Respiratory Rate, Heart Rate, Saturation of Peripheral Oxygen (SPO2) and chest expansion to see the improvement in the patient.

Interventions - In experimental group - PNF respiration will be given to the neonate in supine position.

In control group - No intervention will be given in control group. Outcome measure will be measured at baseline after 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Neonates within eight days of birth Neonates born before 37 weeks of gestation Neonates diagnosed with Respiratory distress syndrome

Exclusion Criteria:

* Medically unstable neonates Neonates who undergone recent surgery or congenital disorder

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-09-02 (Estimated); Primary Completion 2021-01-05 (Estimated); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
Respiratory Rate (RR) | Change in RR measured between baseline and 5th day post intervention
  RR will be assessed from the monitor display (On 1st day prior to intervention and on the 5th day after intervention)
Heart Rate (HR) | Change in HR measured between baseline and 5th day post intervention
  HR will be assessed from the monitor display (On 1st day prior to intervention and on the 5th day after intervention)
Saturation of Peripheral Oxygen (SPO2) | Change in SPO2 measured between baseline and 5th day post intervention
  SPO2 will be assessed from the monitor display (On 1st day prior to intervention and on the 5th day after intervention)
Chest Expansion (CE) | Change in CE measured between baseline and 5th day post intervention
  CE will be measured with the help of measuring tape at nipple level (On 1st day prior to intervention and on the 5th day after intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Saumya Kothiyal, MPT, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Neonatal Intensive Care Unit, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish in scopus or pubmed journal
Supporting Information: Study Protocol, SAP
Time Frame: After ethical approval
Access Criteria: In publically accessible free protocol registration and result system